CLINICAL TRIAL: NCT01810848
Title: Pilot Study of the Impact of Viscosupplementation Therapy With Hylan G-F 20 (Single Injection) on Exercise Tolerance - Implications for Patients With Cardiovascular Risk
Brief Title: Pilot Study of Therapy With Hylan G-F 20 Exercise Capacity
Acronym: CORT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment too low.
Sponsor: OhioHealth (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CORT
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2015-03

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Osteoarthritis; Synvisc; Hylan G-F 20; Exercise; Cardiovascular risk; Knee pain; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hylan G-F 20 (Active Comparator): Patients will receive a single injection of hylan G-F 20 6ml into affected knee. Injections will be performed under fluoroscopic guidance.
  Interventions: Device: Hylan G-F 20
- Control (Sham Comparator): Patients will receive a single sham puncture into the affected knee. Sham punctures will be identical to the treatment injections in all other respects, including duration, use of sterile drapes, sterile preparation, and dimming of the lights. This procedure will include a 22g needle stick through the skin without violating the joint capsule or performing arthrocentesis.
  Interventions: Other: Control

INTERVENTIONS:
Device: Hylan G-F 20 — Synvisc is an elastoviscous high molecular weight fluid which is injected into the knee joint ("intra-articular") for relief of pain from osteoarthritis in patients who have failed to respond adequately to conservative non-pharmacologic therapy and simple analgesics.
  Other Names: Synvisc; Sodium hyaluronate
  Arms: Hylan G-F 20
Other: Control — Control is puncture of the skin at the site of the knee.
  Arms: Control

SUMMARY:
Osteoarthritis of the knee is a degenerative joint disease that involves degradation of the joint. Symptoms include joint tenderness, pain, stiffness, locking, and occasionally an effusion. Over 40 million Americans also have cardiovascular disease in addition to their OA. Initiation and maintenance of even low-levels of physical activity is critical for management of cardiac risk. Patients with osteoarthritis have been shown to have poorer aerobic conditioning, lower daily physical activity levels and lower self-efficacy for exercise than non-OA cohorts.

It has been established that there exists a consistent gradient across activity groups indicating greater longevity and reduced risk of CHD, CVD, and stroke, in more active individuals. Available research suggests the greatest gains in cardiovascular fitness occur in moving a sedentary individual to even low levels of physical activity, and 12 weeks is enough to demonstrate change in the risk profile of at-risk individuals.

Finally, appropriate levels of aerobic and strength training have been shown to be beneficial in treatment of osteoarthritis of the knee. This study will evaluate the effectiveness of hylan G-F 20 (single injection preparation) in promoting greater levels of physical activity and fitness as measured by MET level compared to an exercise-only cohort; evaluating both the change in physical function as well as the cardiovascular risk profile. This is a randomized, single-blinded clinical trial comparing injection of the knee joint with Hylan GF-20 to sham procedure. Subjects will undergo a regular exercise program for 6 months following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals aged between 40 and 70 meeting the American College of Rheumatology (ACR) criteria for primary knee OA with radiographic and symptomatic evidence of TF OA for ≥6 months.
* Radiographic osteoarthritis Kellgren-Lawrence Grade II-III (radiographs taken at entry) in affected knee.
* Average pain numeric rating (defined as moderate level) of 4 - 8 on a scale of zero to 10 over the past week.
* No previous viscosupplement therapy in any joint in past 12 months at the time of randomization.
* No intra-articular steroids in the past 6 months.
* Currently sedentary per American College of Sports Medicine (ACSM) criteria (MET level <9) and at least one of the following cardiovascular risk factors:
* Obesity (BMI between 30 and 40)
* Diabetes mellitus
* HTN (JNC guidelines for HTN stage 1: Systolic >/=140 and diastolic >/= 90)
* Dyslipidemia (ATP3 Guidelines for dyslipidemia: LDL>160, total cholesterol >/=240 and HDL<40)
* Established CAD per clinical or imaging diagnosis
* Allowed medications include stable prescription dose of NSAIDS and/or tramadol. Ad lib use of OTC analgesics will be allowed in both groups.

Exclusion Criteria:

* Grade I and IV OA.
* History of viscosupplementation in any joint in the past 12 months at the time of baseline visit.
* Isolated patello-femoral OA or isolated anterior knee pain (patello-femoral OA co-existing with tibia femoral KOA may be included).
* Symptomatic bilateral knee OA (unless the contra-lateral knee involvement is limited to radiographic OA and not symptomatic).
* Ipsi-lateral symptomatic OA of hip or ankle; contra-lateral symptomatic OA of hip, knee, or ankle, or clinical evidence of hip disease.
* Clinically apparent tense effusion or other acute inflammation of the target knee at baseline.
* History of:

  * Septic OA of any joint
  * Inflammatory arthropathy such as rheumatoid arthritis, gout, pseudogout, lupus, crystalline arthropathy, chondrocalcinosis and other rheumatology diagnosis in judgment of the investigator.
* Active infection of lower extremity (e.g., cellulitis).
* Prosthetic implant in hip and/or lower extremities.
* Any clinical indication for arthroscopic surgery at the time of enrollment.
* Planned surgeries during the trial period (e.g., scheduled/awaiting for arthroscopy or a knee replacement procedure for OA of the knee).
* Plans to initiate other OA treatments including, but not limited to non-pharmacologic, pharmacologic, surgical, chiropractic, acupuncture, yoga, Tai chi, physical therapy during the study period
* Any other intra-articular knee joint injection during the study.
* History of systemic and/or intra-articular steroid injection in target knee within six months of baseline visit.
* History of arthroscopic surgery in affected knee in past 12 months at baseline visit.
* Cruciate/collateral knee ligament instability, ligament laxity, or meniscal instability of target knee.
* Significant alignment deformity such as varus/valgus of target knee in the judgment of the investigator.
* Venous or lymphatic stasis in either leg.
* Peripheral vascular disease.
* Concurrent multi-system or multi-limb trauma.
* Pregnancy or mothers who are breastfeeding. Urine pregnancy test will be administered at baseline for women of childbearing potential.
* On chronic opioid analgesic therapy that cannot be altered. Chronic is defined as ≥6 months.
* Known contraindication to acetaminophen.
* Currently enrolled in another clinical trial or history of trial enrollment within three months at baseline.
* Plans to move/relocate significantly out of area during study period.
* Workman's Compensation beneficiary at base line visit.
* The presence of secondary diagnosis such as neuropathy (any type), radiculopathy, or other nervous system conditions in the judgment of the investigator, contributing to other lower extremity pain that limits activity.
* Physical Therapy for OA of the lower extremity within 6 months prior to enrollment into the study.
* Any musculoskeletal condition besides OA of the knee that limits exercise or normal daily function.
* Acute coronary conditions that are deemed inappropriate for participating in an exercise program.
* Pulmonary conditions limiting functional capacity.
* Known allergy to hylan G-F 20 or any, of its components, or to avian proteins, eggs, feathers, down or poultry.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
MET Level (Exercise capacity) | 6 Months

SECONDARY OUTCOMES:
KOOS (Knee Injury and Osteoarthritis Outcome Score) | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Ruane, DO, Principal Investigator — OhioHealth
Locations (1):
- McConnell Heart Health Center, Columbus, Ohio, United States